CLINICAL TRIAL: NCT03409380
Title: Supplementation Trial on Arginine With Metabolic Profiling
Acronym: STAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Jennifer C. Rood (Unknown); Robbie A. Beyl (Unknown); Martin, Corby, K., M.D. (Individual); Frank L. Greenway (Unknown)
Responsible Party: Principal Investigator, John Apolzan, Asst Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PBRC 2017-027
Record Dates: First submitted 2018-01-11; First posted 2018-01-24 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Protein; Amino Acid; Arginine
Keywords: growth hormone

STUDY DESIGN:
Intervention Model Description: double - blind randomized, crossover design trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arginine (Experimental): Arginine drink provided 1 time. There is about 10 g of arginine in the product.
  Interventions: Dietary Supplement: Arginine Drink
- Placebo (Placebo Comparator): Placebo drink provided 1 time.
  Interventions: Dietary Supplement: Plain Drink

INTERVENTIONS:
Dietary Supplement: Arginine Drink — 10 g of arginine in a formulated drink
  Arms: Arginine
Dietary Supplement: Plain Drink — formulated drink
  Arms: Placebo

SUMMARY:
This study will assess effects of an acute dose of the amino acid arginine on metabolism in healthy young men.

DETAILED DESCRIPTION:
A double - blind randomized, crossover design trial examining arginine vs. placebo beverage treatments will be performed. The primary objective is to determine the effects of arginine assessed by standard laboratory assays and metabolomics. To accomplish the objective standardized meals will be provided for 2 days preceding treatment for dietary consistency. Participants will arrive at the center following a 10-12 hr fast. Blood samples will be collected at baseline (fasting), 1.5 hrs, 3.0 hrs, 6.0 hrs, and 24 hrs post treatment. Plasma prolactin, growth hormone, amino acids, glucose, insulin, triacylglycerols, thyroid hormones (TSH, T3, and T4), sex hormone binding globulin (SHBH), testosterone, cortisol, DHEA, and citrulline will be measured. Metabolomics will be measured at 3 time points for each treatment. Peripheral arterial tonometry (PAT) will also be performed at ~2 hrs following treatment to examine endothelial function in response to nitrous oxide release. In addition, psychological status including fatigue will be assessed using a standardized mood questionnaire (POMS).

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 25 kg/m2.
* Must be physically active (exercise at least 2 days/week).
* Willing to refrain from alcohol and supplements for the duration of the study.
* Willing to refrain from supplement ingestion, nuts, watermelon, and cracklins (fatback) for the 2 weeks prior to the initial treatment diet through the duration of the study.

Exclusion Criteria:

* HIV or AIDS
* Uncontrolled CVD/arrhythmia
* Type I or type II diabetes
* Pregnancy (or breastfeeding)
* Diagnosed eating disorder
* Non-normal sleeping patterns
* Chronic neurological condition
* Altered metabolism including growth hormone disorders
* Use of nicotine or tobacco products
* Heavy caffeine use (≥ 350 mg caffeine/d)
* Whole blood donation within previous eight weeks
* Protein supplementation
* Protein wasting disease.
* Exclusionary medications include diuretics, beta-blockers, weight loss medications or diet pills, anti-inflammatory drugs (corticosteroid/ anabolic steroid/NSAID), antipsychotic medication or other medication that may affect fluid balance, metabolism, or body weight.
* Prisoners and adults who are unable to consent will be excluded from the study.
* Lastly any other medical, psychiatric, or behavioral factors in the judgement of the Principle Investigator that may interfere with study participation or the ability to follow the protocol.

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Growth Hormone | baseline (fasting), 1.5, 3.0, 6.0, and 24.0 hrs
  Change in GH

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No